CLINICAL TRIAL: NCT05078294
Title: Results in Real Clinical Practice of Treatment With Patients With Moderate-severe Atopic Dermatitis
Brief Title: Results in Real Clinical Practice of Treatment of Moderate-severe Atopic Dermatitis
Acronym: Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-DER-2021-01
Record Dates: First submitted 2021-09-09; First posted 2021-10-14 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-09

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients treated as monotherapy with phototherapy, cyclosporine, methotrexate, azathioprine, mycophenolate, dupilumab, baricitinib, upadacitinib, or tralokilumab for the treatment of moderate to severe atopic dermatitis.

SUMMARY:
The purpose of this study is to determine the efficacy results in terms of percentage improvement of the Eczema Area and Severity Index (EASI) as well as on the scale Patient Global Assessment (PGA) throughout the follow-up of patients undergoing subjected to systemic and/or biological treatments in conditions of usual clinical practice. Likewise, collect safety data, recording adverse events related to medication.

DETAILED DESCRIPTION:
This is an observacional follow-up study, open-label (all people know the identity of the intervention), prospective (study following participants forward in time), multi-center study in adult participants with moderate to severe atopic dermatitis. A registration can also be made retrospective data from the patient's medical history.

Participants will be treated with one of this therapy (phototherapy, cyclosporine, methotrexate, azathioprine, mycophenolate, dupilumab, baricitinib, upadacitinib or tralokilumab).

A series of variables will be measured (basal surface area affected (BSA), Eczema Area and Severity Index (EASI), numbers of shoots, analytical determinations and current treatment and adverse effects occurred) in order to observe the changes in the improvement of the disease. Questionnaires will also be carried out to analyze whether the drug acts favorably in improving the disease. Questionnaires like Dermatology Life Quality Index (DLQI), Patient Global Assesment (PGA) and Patient Oriented SCOring Atopic Dermatitis (PO-SCORAD).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years.
* Patients treated with any systemic therapy (other than topical therapy) according to criteria clinical and routine clinical practice. Therefore, the treatments included will be: phototherapy, cyclosporine, methotrexate, azathioprine, mycophenolate, dupilumab, baricitinib, upadacitinib and tralokilumab.
* Patients who grant informed consent.

Exclusion Criteria:

* Patients who do not have the necessary comprehension capacity to understand and sign the informed consent.
* Patients who, according to routine clinical practice, require only topical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population would be patients older than 18 years who suffer from the disease and are being treated with a systemic therapy.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who showed a change in disease severity. | Up to 30 weeks
  Percentage improvement in Eczema Area and Severity Index (EASI) throughout the follow-up of patients undergoing systemic treatments and/or biological.

SECONDARY OUTCOMES:
Medication-related adverse effect rate. | Up to 30 weeks
  Number of adverse effects.
Evaluation of quality of life parameters. | Up to 30 weeks
  Completion of the self-administered dermatology quality of life index questionnaire, which measures the quality of life of the patient.
  Numerical variable (range 0-30) obtained from a self-administered questionnaire already validated in Spanish, which measures the quality of life of surveyed, consisting of 10 questions.

CONTACTS AND LOCATIONS:
Overall Officials: José Juan Pereyra Rodríguez, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (7):
- Spain (7):
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital Universitario Puerta Real, Puerto Real, Cádiz
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Sant Pau, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Arnau de Vilanova, Valencia